CLINICAL TRIAL: NCT07257549
Title: Effectiveness of Real-time Non-invasive Localization for Multiple Lung Nodules: a Pilot, Prospective, Randomized Clinical Trial
Brief Title: Real-Time Non-Invasive Localization for Multiple Lung Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Non-invasive localization
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Preoperative localization; lung nodule; lung cancer; Video-assisted thoracic surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive group (Experimental): Real-time non-invasive localization of multiple pulmonary nodules
  Interventions: Procedure: Real-time non-invasive localization
- CT-guided group (Active Comparator): Manual CT-guided percutaneous needle localization of multiple pulmonary nodules
  Interventions: Procedure: Manual needle localization

INTERVENTIONS:
Procedure: Manual needle localization — Manual needle localization involves the traditional technique of percutaneous localization of pulmonary nodules under CT guidance. The procedure is performed by the physician manually guiding the needle based on real-time CT imaging. The physician adjusts the needle position based on visual cues from the CT scan, which may require multiple attempts for accurate localization. After confirming the needle tip's proximity to the target nodule, indocyanine green (ICG) was injected during deep inspiration to mark the nodule for intraoperative fluorescence imaging. The thoracic surgeon completed resection of the pulmonary nodule based on the area delineated by ICG.
  Arms: CT-guided group
Procedure: Real-time non-invasive localization — The patient underwent a CT scan prior to surgery. The acquired CT image data was saved in DICOM format and subsequently imported into software for three-dimensional reconstruction of the lung lobes, blood vessels, and bronchi. During the procedure, an assistant created a three-dimensional lung model on a separate monitor, aligning it roughly with the orientation of the deflated lung observed via thoracoscopy. The thoracic surgeon then completed resection of the pulmonary nodule guided by the surgeon's three-dimensional lung model.
  Arms: Non-invasive group

SUMMARY:
This study compares real-time non-invasive localization and manual CT-guided needle localization for multiple lung nodules under 20 mm. It primarily aims to evaluate the successful resection rate of pulmonary nodules.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-inferiority clinical study designed to evaluate the effectiveness of a real-time non-invasive localization. The study will be conducted between July 2024 and July 2025, involving 40 patients with multiple lung nodules smaller than 20 mm in diameter. Participants will be randomly assigned to receive either CT-guided manual needle localization or real-time non-invasive localization. The primary outcome measure will be the successful resection rate of pulmonary nodules. Secondary outcome measures will include resection margins, changes in operative approach, intraoperative blood loss, operative time, postoperative hospitalization days, the placement of chest tubes, the duration of chest tube placement, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. the maximum diameter of the lesion on CT did not exceed 20 mm;
2. at least two pulmonary nodules identified;
3. pulmonary nodules showed pure ground-glass opacity (GGO) or mixed GGO on imaging;
4. the outer edge of nodules located between 5-20 mm from the nearest pleural surface.

Exclusion Criteria:

1. nodule location obstructed by the scapula, precluding needle access;
2. proximity of the nodule to major blood vessels, defined as within 2 cm;
3. requirement for localization of multiple pulmonary nodules.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The successful resection rate of pulmonary nodules | Day of surgery.
  The proportion of target lung nodules that are successfully localized and completely resected during the operation, with the target lesion identified in the resected specimen and negative surgical margins confirmed on final pathology.

SECONDARY OUTCOMES:
Resection margins | Day of surgery.
  Distance from the nodule to the resection margin
Changes in operative approach | Day of surgery.
  During surgery, the planned approach must be changed when the target nodule cannot be completely resected due to various reasons.
Intraoperative blood loss | Day of surgery.
  Hemorrhage during surgery.
Operative time | Day of surgery.
  Total duration of the thoracic surgical procedure, measured in minutes from skin incision to completion of skin closure for the index operation.
Postoperative hospitalization days | Perioperative.
  The postoperative hospitalization duration refers to the total number of days the patient remains in the hospital from the completion of surgery until discharge.
The placement of chest tubes | Day of surgery.
  Determine whether a chest tube needs to be placed based on the patient's condition during surgery.
The duration of chest tube placement | Perioperative.
  The chest tube placement duration refers to the number of days from the placement of the chest tube after surgery until its removal.
Postoperative complications | Perioperative.
  Postoperative complications refer to any adverse events or symptoms that occur after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated of Guangzhou Medical University, Guangzhou, Guangdong, China